CLINICAL TRIAL: NCT07085325
Title: CSIMEMPHIS: Long-term Follow-up of Medulloblastoma Survivors That Received Craniospinal Irradiation
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CSIMEMPHIS; NCI-2025-07105 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2025-07-02; First posted 2025-07-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Medulloblastoma
Keywords: Medulloblastoma; Survivor
MeSH Terms: conditions — Medulloblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic Testing - Germline genetic studies (whole genome and exome) will be performed and banked specifically for future use by CSIMEMPHIS investigators.
  Gut Microbiome - Stool self-collection will occur around the time of study visits, with samples stored at room temperature in tubes within ziplock bags for up to 24 hours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSIMEMPHIS-only Group: Participants meeting the CSIMEMPHIS eligibility criteria.
- BRAINatomy2 Group: In addition to meeting the eligibility criteria for CSIMEMPHIS, the Brainatomy2 cohort participants must be able to tolerate non-sedated MRI and must not have a history of clinically significant PFS.

SUMMARY:
The study is being done to learn more about the long-term health and well-being of participants treated for medulloblastoma. The study is to decide which evaluations focusing on therapy-related lasting effects (or toxicities) should be considered.

Medulloblastoma outcomes have improved with contemporary therapies including modern neurosurgical techniques and risk-adapted radiotherapy and chemotherapy regimens. However, survivors remain at risk for long-term health problems such as neurocognitive deficits, hearing loss, impaired cardiorespiratory fitness and physical performance, cardiac and neuroendocrine dysfunction, musculoskeletal conditions, and infertility.

DETAILED DESCRIPTION:
This is initially a cross-sectional timepoint serving as the baseline for prospective follow-up to evaluate health outcomes in a population of childhood medulloblastoma survivors treated with contemporary therapy, including both photon and proton Craniospinal irradiation (CSI).

Participants will be invited to enroll on both SJLIFE and this protocol. This study will utilize the St. Jude Lifetime Cohort (SJLIFE) infrastructure to comprehensively evaluate 5-year survivors of childhood medulloblastoma treated with radiation therapy on or according to SJMB12, including those treated with differing doses and modalities of CSI. Insights gained on late effects will inform long-term surveillance and may identify novel outcomes, guiding future studies. Participants and their parents/guardians will also be asked to complete surveys that assess patient-reported outcomes.

There will be two cohorts of participants - CSIMEMPHIS (all participants who meet initial eligibility criteria) and BRAINatomy2. To be eligible for the Brainatomy2 cohort, survivors must be able to tolerate non-sedated MRI and must not have a history of clinically significant PFS. Recruitment of these patients will be led by staff in Radiation Oncology.

All study participants undergo the SJLIFE comprehensive set of medical evaluations that target overall health and function as well as possible treatment-related toxicities. CSIMEMPHIS participants will undergo testing tailored to medulloblastoma treatment and follow-up. All participants will undergo fMRI at the CSIMEMPHIS visit. For those eligible for BRAINatomy2, the BRAINatomy2 investigational fMRI will be prioritized and all others will undergo the CSIMEMPHIS investigational fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any subtype of medulloblastoma between the ages of 3 to 22 years or between the ages of 22 to 44 years with the sonic hedgehog (SHH) subtype of medulloblastoma
* Radiotherapy on or according to the SJMB12 protocol
* 5 or more years since the initiation of radiation therapy and who did not have evidence of disease progression
* Provision of informed consent by participant/guardian or legal representative; Assent by minor participant
* Participants may choose to complete all or a subset of the proposed assessments; refusal to participate in some aspects of the study will not preclude participant inclusion
* Participants must also complete enrollment on SJLIFE

Exclusion Criteria:

* Participants or their legal guardian/representative are unwilling or unable to provide written informed consent.
* Participants who had relapsed or refractory disease during or following completion of treatment for medulloblastoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
To describe and compare the long-term health outcomes among medulloblastoma survivors treated with radiation therapy on or according to the SJMB12 protocol with varying craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  In the SJLIFE study Survivors will undergo the SJLIFE core battery of testing with a focus on outcomes for which early evidence has demonstrated the potential association between proton therapy and reduced late-effect burden. Testing includes neuromuscular function, laboratory testing, neurocognitive assessments, physiologic assessments, and outcome questionnaires.

SECONDARY OUTCOMES:
To correlate the spatial distribution of radiation dose with neurologic, endocrine, cognitive, and physiologic outcomes among a subset of medulloblastoma survivors, using both conventional and voxel-based analysis. | Baseline
  Subjects selected for the Brainatomy2 study will undergo a one-time investigational MRI/fMRI study designed to target working memory and processing speed. The investigational MRI/fMRI exam includes Axial T2 weighted imaging for post-surgical and post-radiotherapy assessment of brain parenchymal changes, and 3D isometric voxel T1 volume imaging for structural analysis of the whole brain. It also employs pulsed ASL technique for voxel-based cerebral blood flow assessment and diffusion imaging to generate ADC and FA maps, normalizing anatomical connectivity maps to the T1 volume. Additionally, resting-state functional MRI (fMRI) provides whole brain coverage for analyzing temporal co-activation in BOLD fMRI maps in relation to cognitive testing results.

OTHER OUTCOMES:
Analyze regional differences in brain activity using fMRI among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens and radiation modalities. | Baseline
  Subjects selected for Brainatomy2 will undergo a one-time investigational MRI/fMRI exam for post-surgical and post-radiotherapy assessment of brain parenchymal changes, and structural analysis of the whole brain. The exploratory endpoints focus on imaging assessments: Perfusion imaging with median regional cerebral blood flow map registration to T1 MPRAGE structural brain imaging, Diffusion and Diffusion Tensor Imaging with median Apparent Diffusion Coefficient map registration to structural brain imaging, including the generation of whole-brain anatomic connectivity maps, and Resting state fMRI with whole brain coverage, analyzing differences in functional connectivity between processing speed groups through voxel-by-voxel comparisons.
To investigate the long-term impact of posterior fossa syndrome among medulloblastoma survivors including neurological brain activity with cognitive function. | Baseline
  fMRI maps brain activity associated with cognitive functions such as memory, attention, language, and executive function. It can reveal patterns of brain reorganization corresponding with cognitive test scores and declines in performance. By integrating fMRI findings with cognitive testing and other measures, we can study differences in treatment such as craniospinal dose and better understand the neural mechanisms underlying cognitive disorders and related complications. fMRI findings can be mapped to the spatial distribution of radiation dose using conventional and voxel-based analysis.
To investigate the long-term impact of posterior fossa syndrome among medulloblastoma survivors including speech and language. | Baseline
  To determine impact of speech and language, hearing is evaluated with tympanometry, pure-tone audiometry at 250, 500, 1000, 2000, 3000, 4000, 6000, and 8000 Hz, and speech audiometry in quiet. Speech-in-noise tests measure the ability to hear and understand speech in background noise.
To assess health-related quality of life (HRQOL) among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  We will utilize these instruments in addition to the SJLIFE Comprehensive Health Form to evaluate quality of life. This 23-item questionnaire encompasses physical functioning, emotional functioning, social functioning, and school functioning. Items are scored to create a Psychosocial Health Summary Score (0 to 100 scale), with a higher score indicating better health-related quality of life (HRQOL). Self-report measures are available for children and adolescents aged 5 to 18 years, and parent proxy-report measures are available for those aged 2 to 18 years.
To map changes in the working memory structural connectome among medulloblastoma survivors treated with varying craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Subjects will be given processing speed tasks performed together while in the scanner. The N-back task, they are required to respond, using the response button, when they see the same stimulus repeated after N intervening stimuli. The stimuli used will be line drawings of everyday objects. The task will last 5 minutes. Object snap task and Silly sentence task are two processing speed tasks using pictures and sentences. For the Object snap task, they are required to respond yes when two object pictures, presented at the same time, are identical. Subjects are required to respond quickly, but accurately. The fMRI paradigm will use NordicNeuro Lab software.
To explore the association of social drivers of health (SDOH) with health outcomes among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  This will be evaluated using the Family Environment Scale to assess the environmental characteristics of the family. A Brief Symptom Inventory-18 will be administered to measure parental/caregiver emotional distress. The Parent Protection Scale will be administered to evaluate parental protective behavior. The census tract-based Social Vulnerability Index (SVI) will be used to evaluate neighborhood adversity per the patient's residential address. Collectively these surveys will show interplay between socioeconomic status and environmental factors that influence health outcome disparities.
To evaluate and compare the neurologic effects, complications, surgical injury, and second neoplasms among medulloblastoma survivors treated with varying craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Sleep will be assessed to determine the effects from surgery, treatment, and complications using polysomnography evaluation and various sleep surveys assessing quality of sleep, sleep patterns, drowsiness during the day, and insomnia.
To examine and compare endocrinologic effects and complications, including fertility, among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  The following lab measures will be collected LH, AMH, FSH, inhibin B, and testosterone in males aged ≥ 9 years and LH, FSH, estradiol, and AMH in females aged ≥ 8 years. Additional endocrine lab assessments will include hemoglobin A1c, insulin, lipid panel, vitamin D 25-OH, morning cortisol, IGF-1, TSH, and free T4. Tanner staging will be performed as part of the clinical exam regardless of age until fully developed (Tanner stage 5). A bone radiograph will be obtained for participants < 18 to assess skeletal maturation in relation to chronological age to assess growth and pubertal development. Thyroid ultrasound will assess thyroid nodules. Dual x-ray absorptiometry (DXA) scan obtained will be used to estimate total and specific regional relative lean mass values, visceral fat, subcutaneous adipose tissue, and appendicular lean mass.
To characterize and compare cognitive effects among medulloblastoma survivors treated with varying craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Neurocognitive outcomes will be evaluated with age-appropriate measures using a battery of standardized tests. The core battery of cognitive tests will ensure that long-term neurocognitive and learning sequelae of treatment are captured.
To evaluate and compare physiologic effects and complications (cardiorespiratory) among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Electrocardiogram will be used to evaluate for rhythm and conduction abnormalities. Pulmonary function will be measured with pulmonary function tests (PFTs). For patients under 5 years of age or those that cannot perform adequate testing, pulse oximetry will be the primary measure of pulmonary function. Cardiorespiratory fitness will be evaluated with maximal cardiopulmonary exercise testing (CPET) on a treadmill using a modified Bruce protocol, or with an arm or leg ergometer for participants with impairments that prohibit walking on a treadmill. Heart Rate Variability (HRV) will be assessed remotely using photoplethysmogram (PPG) data collected using the LEAP® wrist biosensor. Stool self-collection will occur and overall diversity and microbiome compositional attributes will be compared.
To evaluate and compare physiologic effects and complications (gut microbiome) among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Stool self-collection will occur, and composition will be assessed using DNA extracted from frozen aliquots. The extraction will be conducted using the Chemagic 360 system, followed by 16S rRNA gene amplification by touchdown PCR and sequencing at St Jude Hartwell Center. Overall diversity and microbiome compositional attributes will be compared.
To evaluate and compare physiologic effects and complications (musculoskeletal) among medulloblastoma survivors treated with different craniospinal doses, chemotherapy regimens, and radiation modalities. | Baseline
  Growth velocity, the change in height and weight over time, is a more sensitive measure of growth than a single height or weight. Spinal MRI of the spine will be used to assess for scoliosis, kyphosis, vertebral body wedging, spinal height loss, degenerative disc, and degenerative bone changes. Sitting height will also be obtained to evaluate for skeletal dysplasia or impaired spinal growth.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Merchant, DO, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols